CLINICAL TRIAL: NCT01326078
Title: Comparison Between Propofol Nanoemulsion and Propofol Lipid Emulsion on Children Undergoing Ambulatory Invasive Procedures.
Brief Title: Use of Lipid Emulsion or Nanoemulsion of Propofol on Children Undergoing Ambulatory Invasive Procedures.
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The Sponsor has no interest in continuing the study.
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Collaborators: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CRIST011
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Leukemia
Keywords: sedation; children; leukemia; bone marrow biopsy
MeSH Terms: conditions — Leukemia | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol nanoemulsion (Experimental): 3-4 mg/kg of propofol nanoemulsion will be administered by 1mL per 5 seconds, adjustment dose can be given.
  Interventions: Drug: propofol
- propofol lipid emulsion (Active Comparator): 3-4 mg/kg will be administered by 1 ml per 5 seconds.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — 3 - 4 mg/kg IV, adjustment dose if necessary

SUMMARY:
The purpose of this study is to compare the safety and efficacy of the of propofol nanoemulsion and lipid emulsion for sedation in non-invasive ambulatory procedures.

DETAILED DESCRIPTION:
Nanoemulsion of propofol has been developed without lipid solvent in the formulation to minimize the adverse events such as pain of injection, redness, heat, phlebitis.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar Puncture or Myelogram
* Peripheral Intravenous access available in the veins on the dorsal region of the hand
* The informed consent signed by the legal responsible of the child allowing the participation in the study

Exclusion Criteria:

* Relative or absolute contraindications use of propofol and excipients
* Contraindications to the patient undergo general anesthesia or sedation with drug
* Allergy derived from egg or soy
* Use of pre-medication
* Patient receiving psychotropic drugs
* Use of opioid within 24 hours
* The responsible for the children unable to decide for his participation
* The severity of the condition wich compromises vital functions such as ventilation and hemodynamic balance
* Liver cancer which compromises its function
* Changes in the blood tests
* Others comorbidities in the investigator opinion

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Classification of the sedation level | time 0
  Instantly after the loss of consciousness (loss of corneal-palpebral reflex) will be measured the sedation using the Ramsay Modified Scale.

SECONDARY OUTCOMES:
Time of latency | 3-10 seconds
  Time between the injection and loss of the corneal-palpebral reflex
Pain at injection | 3 - 10 seconds: during the injection
  The pain will be measured by CHEOPS Scale which evaluates the behavior of the child against pain.
Physician satisfaction | 12 hours: end of procedure
  The satisfaction of the medical specialist will be assessed through a questionnaire that assesses conditions of sedation for the procedure.
Awakening time | 10 hours: when the patient awakes
  Time between the last dose of propofol and the time when the patient awakes (cry, eyes opening and spontaneous movement).
Total dose | 12 - hours End of procedure
  The total dose used will be measured in mg/kg/hour.
Incidence of Adverse Events | 0 to 14 hours
  Adverse events will be compared in its incidence in the two formulations of propofol during the anesthetic induction and 12 hours after the procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana C Lima, PhD, Principal Investigator — IMIP